CLINICAL TRIAL: NCT07259226
Title: International Multicenter Multicohort Open-label Phase II Trial Aiming to Define Optimal Methods for Predicting Response/Resistance to Antibody-drug Conjugates in Patients With Solid Tumors Treated According to Current Standard Indications.
Brief Title: Optimal Methods to Characterize ADC Resistance in Solid Tumors and Identify Clinically Useful Biomarkers
Acronym: OASIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UC-TRA-2507; ID RCB 2025-A01462-47 (Other: ANSM)
Record Dates: First submitted 2025-09-26; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced Breast Cancer; Advanced Gastric Cancer; Advanced Urothelial Cancer; Advanced Non Small Cell Lung Cancer (NSCLC)
Keywords: ADC; resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T-DXd (trastuzumab deruxtecan) (Other): Standard of care T-DXd indication
  Interventions: Procedure: Biological samples collection; Behavioral: questionnaires to collect patient reported outcomes
- T-DM1 (trastuzumab emtansine) (Other): Standard of care T-DM1 indication
  Interventions: Procedure: Biological samples collection; Behavioral: questionnaires to collect patient reported outcomes
- SG (sacituzumab govitecan) (Other): Standard of care SG indication
  Interventions: Procedure: Biological samples collection; Behavioral: questionnaires to collect patient reported outcomes
- EV (enfortumab vedotin) (Other): Standard of care EV indication
  Interventions: Procedure: Biological samples collection; Behavioral: questionnaires to collect patient reported outcomes

INTERVENTIONS:
Procedure: Biological samples collection — Biological samples collection (tumor tissue, blood, sputum) before initiation of treatment, during treatment, and at treatment discontinuation.
  Other Names: Blood sample collection; Sputum sample collection; Tumor tissue sample collection
Behavioral: questionnaires to collect patient reported outcomes — QLQ-C30, QLQ-FA12, HADS, EQ-5D 5L

SUMMARY:
International study that will evaluate the association of prespecified biomarkers with resistance to Antibody-drug conjugates (ADCs), a type of targeted cancer treatment currently used in clinical practice for treating different tumor types.

DETAILED DESCRIPTION:
Over the past five years, antibody-drug conjugates (ADCs) have dramatically improved survival in solid and hematologic malignancies. Among 14 ADCs approved worldwide, nine are now available in Europe, and over 370 others are in clinical development. This expanding landscape indicates that ADCs could soon replace conventional chemotherapy across multiple tumor types. Given this rapid evolution, clinicians will need to select the most suitable ADC for each patient, considering tumor biology, microenvironment (TME) and patient-specific factors. Yet, despite remarkable efficacy, resistance to ADCs eventually arises. Understanding resistance mechanisms is therefore essential to guide therapeutic sequencing and optimize next-generation ADCs.

ADCs are complex molecules combining an antibody, a linker, and a cytotoxic payload. Their activity depends on factors such as antigen expression, internalization, linker stability, and payload sensitivity. Resistance can result from altered vascular perfusion, antigen downregulation, defective internalization or trafficking, impaired linker cleavage, drug efflux, or payload target modifications. These multifactorial processes differ from those driving resistance to traditional chemotherapies. Existing preclinical and clinical tools (Patient-Derived Xenograft(PDX)/Cell-line-Derived Xenograft (CDX) models, standard imaging, Immunohistochemistry (IHC), genomic profiling) fail to capture this complexity or predict ADC efficacy and resistance. Furthermore, ADCs often cause significant toxicities-on-target or off-target-affecting the ocular surface, skin, lungs, and peripheral nerves. Patient factors such as age, comorbidities, and weight influence these events. Understanding the determinants of toxicity is critical to maintain quality of life and treatment adherence.

The OASIS program aims to identify predictive biomarkers of ADC response and toxicity to enable personalized ADC selection and toxicity prevention. This multicenter study will integrate advanced technologies-digital pathology, liquid biopsy, and Patient-derived organoids (PDOs)-to generate comprehensive biological and clinical data. Using these datasets, a multimodal machine-learning model (OASIS Multiparametric Score) will be developed to predict both efficacy and key toxicities of ADCs. The project will prospectively include patients receiving ADCs in standard practice, with longitudinal tumor and blood sampling to investigate biomarkers of resistance and toxicity. In parallel, preclinical models derived from patient tumors will explore resistance mechanisms and screen ADC sensitivity.

A retrospective cohort of patients previously treated with ADCs will first be analyzed to prioritize biomarker candidates based on published data and prior findings. From this, five binary biomarkers will be selected for the primary objective. Combined with prospective data, this retrospective work will expand the translational biobank and support the construction of the OASIS score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed a written informed consent form prior to any trial specific procedures;
2. Patients must be ≥18 years old;
3. Histologically confirmed or radiologically documented unresectable locally advanced or metastatic cancer (Breast, Urothelial, Non small Cell Lung or Gastric) with an indication to receive an Antibody-Drug Conjugate (ADC) approved or accessible through an early access program;
4. Patients must have at least 2 tumor lesions (primary tumor can be included): at least one measurable tumor lesion for tumor evaluation according to response evaluation criteria in solid tumors (RECIST) V1.1 and at least one tumor lesion other than bone and brain for biopsy;
5. Patients must have a metastatic or locally advanced tumor site easily accessible to biopsy (with exception of bone and brain metastasis) and must have agreed to perform pretreatment and post-treatment biopsies; an archival pre-treatment biopsy may be used if it was collected within one month of enrolment, if no anticancer therapy was administered after the biopsy and if sufficient material is available for research;
6. Life expectancy must be ≥12 weeks according to the discretion of the investigator;
7. ECOG performance status ≤ 2;
8. Patients must have adequate hematologic and organ function, compatible with ADC administration, as per drug-specific recommendations;
9. Women of childbearing potential and male patient must agree to use adequate contraception for the duration of trial participation and up to 7 months after completing treatment for women and up to 4 months for men;
10. Patients must be affiliated to a social security system (or equivalent);
11. Patients must be willing and able to comply with the protocol for the duration of the trial;
12. Patients must consent to the use of their collected tumor specimen, as well as, blood samples as detailed in the protocol for future scientific research, which includes but is not limited to DNA, RNA, and protein-based biomarker analysis.

Exclusion Criteria:

1. Patients treated with an antibody drug conjugate in a curative setting;
2. Patients who did not consent to sample use;
3. Presence of another progressive pathology with short-term life-threatening prognosis;
4. Patients undergoing concurrent treatment for a malignancy or hematologic disorder distinct from the indication for which the ADC is being administered.
5. Patients with inadequate washout period prior to Cycle 1 Day 1, defined as:

   * Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days.
   * Any cytotoxic chemotherapy, investigational agents or other anticancer drug(s) (including another ADC) from a previous cancer treatment regimen or clinical study (other than epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI)), <14 days or 5 half-lives, whichever is longer.
   * Immune checkpoint inhibitor therapy <21 days.
   * Hormonal therapy <21 days.
   * Major surgery (excluding placement of vascular access) <28 days.
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <14 days.
6. Female participant who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 90 days after the final administration of study treatment;
7. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of resistance to ADC | Through study completion, an average of 3 years
  Resistance is defined by differences in the frequency (higher or lower) of molecular aberrations detected between paired baseline samples and progression samples (i.e., samples collected at the time of disease progression under ADC treatment)

SECONDARY OUTCOMES:
Additional biomarkers of resistance characterised by histology | Through study completion, an average of 3 years
  Differences in the frequency of molecular aberrations characterised by histologic/proteomic/genomic/transcriptomic analysis between samples of patients progressing on ADC and paired pre-treatment samples (beyond biomarkers of primary outcome)
Biomarkers of ADC outcome | From first day of cycle 1 (each cycle is 21 to 28 days) to date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-Free Survival (PFS) defined as the time from start of treatment and radiological progression or death, whichever occurs first. Tumor assessments are made by local investigators as per standard practice (RECIST 1.1.). Patients still alive at the cut-off time without documented progression (including lost to follow-up) will be censored at the time of latest evaluable efficacy assessment.
Biomarkers of ADC outcome | From first day of cycle 1 (each cycle is 21 to 28 days) to date of 6 months of treatment completion
  Objective Response Rate (ORR) defined as the proportion of patients with a confirmed complete response (CR) or partial response (PR) assessed by investigators after 6 months of treatment.
Biomarkers of ADC outcome | From first day of cycle 1 (each cycle is 21 to 28 days) to date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Clinical Benefit Rate (CBR) defined as the proportion of patients who had a CR, PR, or stable disease for 6 months or more.
Biomarkers of resistance to ADC | From first day of cycle 1 (each cycle is 21 to 28 days) to date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Duration of response (DOR) defined as the time from treatment initiation to disease progression or death for patients who achieve CR or PR.
Biomarkers of ADC outcome | From first day of cycle 1 (each cycle is 21 to 28 days) to date of death from any cause, assessed up to 60 months
  Overall Survival (OS) defined as the time from inclusion to death due to any cause. Patients still alive at the cut-off time (including lost to follow-up) will be censored at the last known alive date.
Expression of ADC target measured on CTC and within tumor tissue | Through study completion, an average of 3 years
  Concordance between ADC target expression (HER2, TROP-2, Nectin-4) on pre- and post-treatment tumor biopsy (IHC) and antigen expression on Circulating Tumor Cells (CTCs).
Patients' reported outcomes (PROs) | Through study completion, an average of 3 years
  Overall quality of life will be assessed using the EORTC-QLQ-C30 and EQ-5D-5L at Baseline, after 3 months of treatment completion, at treatment discontinuation (for progression or any other reason)
Patients' reported outcomes (PROs) | Through study completion, an average of 3 years
  Fatigue will be assessed using QLQ-FA12 at Baseline, after 3 months of treatment completion, at treatment discontinuation (for progression or any other reason).
Patients' reported outcomes (PROs) | Through study completion, an average of 3 years
  Anxiety and depression will be assessed using HADS questionnaire at Baseline, after 3 months of treatment completion, at treatment discontinuation (for progression or any other reason)
Treatment cost | Through study completion, an average of 3 years
  Number of resources consumed in terms of treatment, hospitalization (for drug administration and toxicity), biological and radiological exams during the ADC treatment, in order to calculated the corresponding management cost.
ADC-related specific toxicities | Through study completion, an average of 3 years
  Safety as measured by the frequency and severity of key ADC toxicity (Interstitial Lung Disease, skin toxicity, ocular toxicity, peripheral neuropathy) as measured by NCI-CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pistilli, MD, PhD, Principal Investigator — Gustave Roussy Cancer Center
Locations (1):
- Gustave Roussy Cancer Center, Villejuif, France

IPD SHARING:
Plan to Share IPD: No